CLINICAL TRIAL: NCT06527703
Title: International Prospective, Observational, Multi-centre, Cross-sectional Study on the Duration of Pre-operative Liquid Fasting
Brief Title: An International Prospective, Observational, Multi-centre Study on the Duration of Pre-operative Liquid Fasting
Acronym: THIRST
Status: Completed | Type: Observational
Sponsor: Mater Dei Hospital, Malta (Other)
Collaborators: Puerta de Hierro University Hospital (Other)
Responsible Party: Principal Investigator, Anne Marie Camilleri Podesta', Dr, Mater Dei Hospital, Malta
Other Study IDs: ThirstStudy
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus; Hypertension; Ischaemic Heart Disease; Comorbidities and Coexisting Conditions; Fasting; Fasting, Time Restricted
Keywords: Preoperative fluid fasting time
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Coronary Artery Disease; Fasting; Intermittent Fasting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- preoperative liquid fasting duration in adult patients undergoing elective surgery: Adult patients scheduled for elective procedures and either requiring general anaesthetic, regional anaesthesia or sedation will be eligible to participate. The necessary institutional approvals will be obtained.
  Data will be collected on the same day among the participating centres. After obtaining consent and screening for eligibility, the patients will answer a short questionnaire regarding their last liquid intake.
  The type of procedure, type of anaesthesia and time of arrival in the holding bay / operating room as well as the date and time at which clear fluids were last consumed will be recorded
  Interventions: Other: no intervention
- preoperative liquid fasting time: Adult patients scheduled for elective procedures and either requiring general anaesthetic, regional anaesthesia or sedation will be eligible to participate. The necessary institutional approvals will be obtained.
  Data will be collected on the same day among the participating centres. After obtaining consent and screening for eligibility, the patients will answer a short questionnaire regarding their last liquid intake.
  The type of procedure, type of anaesthesia and time of arrival in the holding bay / operating room as well as the date and time at which clear fluids were last consumed will be recorded
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — Patients have to answer a questionnaire. The following data will be recorded:
  Patient Number:
  Informed Consent: ☐ yes ☐ no
  Screening for eligibility Age >/= 18 years: ☐ yes ☐ no Gender: ☐ M ☐ F Patient undergoing elective procedure: ☐ yes ☐ no
  Time of arrival in the operating room _________________
  Procedure:
  General surgery ☐ Orthopaedic surgery ☐ Neurosurgery ☐ Cardiac surgery ☐ Vascular ☐ Urology ☐ ENT/ dental/ maxillo-facial ☐ Obstetrics and Gynaecology surgery ☐ Ophthalmic surgery ☐ Non-operating room anaesthesia ☐ Endoscopy ☐ Other ____________________
  Type of Anaesthesia (choose 1):
  GA ☐ Sedation ☐ Regional ☐
  Date and Time at which clear fluids were last consumed:_______________________

SUMMARY:
The investigators will be performing an international prospective, observational, multi-centre, cross-sectional study to determine the actual duration of preoperative liquid fasting time in European patients.

Research has shown that prolonged fasting, particularly for liquids, is likely harmful to patients before, during, and after an operation. Harm from prolonged fasting for liquids includes dehydration, dysregulated blood sugar levels, increased stress response, and postoperative complications. Recent studies show an average preoperative fasting time for liquids that are significantly longer than necessary.

Reducing fasting time is associated with improved patient well-being, a smoother perioperative course, shorter hospital stays, cost savings, and enhanced environmental sustainability.

The investigators hypothesize that excessive preoperative fasting is still common practice in most European countries and would like to investigate the actual length of liquid fasting practices amongst patients in Europe, to determine whether the current guidelines are being followed.

DETAILED DESCRIPTION:
The investigators will be performing an international prospective, observational, multi-centre, cross-sectional study to determine the actual duration of preoperative liquid fasting time in European patients. The investigators have interest and commitment from 12 countries and hope to recruit more hospitals in the coming weeks.

Research has shown that prolonged fasting, particularly for liquids, is likely harmful to patients before, during, and after an operation. Harm from prolonged fasting for liquids includes dehydration, dysregulated blood sugar levels, increased stress response, and postoperative complications. Recent studies show an average preoperative fasting time for liquids that are significantly longer than necessary.

In the pilot study the investigators conducted a few weeks ago, the average preoperative liquid fasting time was 12 hours instead of the recommended 2 hours. Reducing fasting time is associated with improved patient well-being, a smoother perioperative course, shorter hospital stays, cost savings, and enhanced environmental sustainability. The investigators hypothesise that excessive preoperative fasting is still common practice in most European countries and would like to investigate the actual length of liquid fasting practices amongst patients in Europe, to determine whether the current guidelines are being followed. This will give further insight to colleagues and encourage healthcare professionals to follow the fasting guidelines from the European Society of Anaesthesia and Intensive Care.

The methodology and other details can be found in the study protocol and the other documents. Adult patients scheduled for elective procedures and either requiring general anaesthetic, regional anaesthesia or sedation will be eligible to participate. Data will be collected on the same day among the participating centres and the target date is the 23rd October 2024.

After obtaining consent and screening for eligibility, the patients will answer a short questionnaire regarding their last liquid intake. The following data will be collected:

Patient Number:

Informed Consent: ☐ yes ☐ no

Screening for eligibility Age >= 18 years: ☐ yes ☐ no

Gender: ☐ M ☐ F Patient undergoing elective procedure: ☐ yes ☐ no Time of arrival in the operating room _________________

Procedure:

General surgery ☐ Orthopaedic surgery ☐ Neurosurgery ☐ Cardiac surgery ☐ Vascular ☐ Urology ☐ ENT/ dental/ maxillo-facial ☐ Obstetrics and Gynaecology surgery ☐ Ophthalmic surgery ☐ Non-operating room anaesthesia ☐ Endoscopy ☐ Other ____________________

Type of Anaesthesia (choose 1):

GA ☐ Sedation ☐ Regional ☐

Date and Time at which clear fluids were last consumed:_______________________

The questionnaire will last less than 5 minutes.

This questionnaire is very simple and no patient identifiable data will be recorded on the data collection tool.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patients undergoing elective surgery
3. Written informed consent

Exclusion Criteria:

1. Age < 18 years
2. Urgent and emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for elective procedures and either requiring general anaesthetic, regional anaesthesia or sedation will be eligible to participate.
  Data will be collected on the same day among the participating centres. After obtaining consent and screening for eligibility, the patients will answer a short questionnaire regarding their last liquid intake.
  The type of procedure, type of anaesthesia and time of arrival in the holding bay / operating room as well as the date and time at which clear fluids were last consumed will be recorded
Sampling Method: Non-Probability Sample
Enrollment: 5100 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
The primary objective of this observational study is to determine the actual duration of preoperative liquid fasting time. | Data will be collected on the same day among the participating centres. This is planned for the 23rd October 2024
  Adult patients scheduled for elective procedures and either requiring general anaesthetic, regional anaesthesia or sedation will be eligible to participate.
  After obtaining consent and screening for eligibility, the patients will answer a short questionnaire regarding their last liquid intake.

CONTACTS AND LOCATIONS:
Overall Officials: Federico Bilotta, Prof, Principal Investigator; Anne Marie Camilleri Podesta, Dr, Principal Investigator — Mater Dei Hospital
Locations (1):
- Mater Dei Hospital, San Ġiljan, Msida, Malta

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD The results from the study will be published

REFERENCES:
- [Derived] Camilleri Podesta AM, Sciberras S, Moisa E, Valletta L, Farrugia S, Paal P, Kouki P, Gasiunaite D, Vide S, Varosyan A, Golubovska I, Durnev V, Chkhaidze M, Kuci S, Vujovic B, Bilotta F. Preoperative liquid fasting practices in twelve European countries: A prospective multicentre cohort study (Thirst study). Eur J Anaesthesiol. 2026 Jan 8. doi: 10.1097/EJA.0000000000002347. Online ahead of print. PMID 41504282